CLINICAL TRIAL: NCT03024541
Title: Longitudinal Analysis of Cumulative Exposure to Anticholinergic and Sedative Drugs Measured With the Drug Burden Index
Brief Title: Longitudinal Analysis of Drug Burden Index
Status: Completed | Type: Observational
Sponsor: University of Groningen (Other)
Responsible Party: Principal Investigator, Katja Taxis, Professor, University of Groningen
Other Study IDs: DBI InterRAI LASA
Record Dates: First submitted 2016-10-18; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Polypharmacy; Anticholinergics; Hypnotics and Sedatives; Cognitive Function; Physical Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- LASA study
- InterRAI consortium

SUMMARY:
Anticholinergic and sedative drugs are frequently prescribed to older people, despite their negative impact on older people's physical and cognitive function. To estimate the cumulative exposure to anticholinergic and sedative drugs, Hilmer et al. published the Drug Burden Index (DBI) in 2007. The present study aims to complement previous study findings showing higher DBI values to be associated with physical and cognitive impairment. Most previously conducted studies of the DBI were either cross-sectional or were longitudinal but with short follow-ups. Furthermore, it remains unknown whether higher DBI values carry extra risks for patients with dementia. Finally, relatively little is known about the stability of DBI values over time. The current project therefore aims to examine (1) longitudinal relationships between long-term cumulative exposure to anticholinergic and sedative drugs as measured with the DBI and cognitive and physical function, (2) to examine interaction effects between DBI exposure and dementia, and (3) to examine trajectories of DBI exposure, i.e. DBI exposure remaining stable, declining, increasing or fluctuating over time. These project aims will be studied with longitudinal data from eligible participants > 60 years from the LASA study with participants being followed-up during two decades, and the longitudinal data from the InterRAI consortium. Various clinical outcomes regarding cognitive and physical function will be studied. Data will be analysed with generalised linear mixed models and Latent Class Growth Analysis.

ELIGIBILITY:
LASA:

Inclusion criteria:

* 55 years and older

Exclusion criteria:

* problem drinkers in the past and the present
* very severe vision and hearing problems

InterRAI:

Inclusion criteria:

* 55 years or older

Exclusion criteria:

* consumption of 5 or more units of alcohol on one occasion
* unknown sex or age

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People aged 55 years and older, both community-dwelling individuals and individuals living in residential aged care facilities
Sampling Method: Probability Sample
Enrollment: 9985 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
LASA study: Alphabet Coding Task | 21 years: 7 waves separated by 3 year intervals

SECONDARY OUTCOMES:
LASA study: Mini Mental Status Examination | 21 years: 7 waves separated by 3 year intervals
LASA study: Verbal Fluency Test: Phonemic fluency | collected at 7th wave after 21 years (cross-sectional)
LASA study: Verbal Fluency Test: Semantic fluency | collected at 7th wave after 21 years (cross-sectional)
LASA study: Digit Span Forward from Wechsler Adult Intelligence Scale | collected at 7th wave after 21 years (cross-sectional)
LASA study: Digit Span Backward from Wechsler Adult Intelligence Scale | collected at 7th wave after 21 years (cross-sectional)
LASA study: 15-Words Test: Word Learning | 21 years: 7 waves separated by 3 year intervals
LASA study: 15-Words Test: Delayed Recall | 21 years: 7 waves separated by 3 year intervals
LASA study: Functional Independence Scale | 18 years: 6 waves with 3 year intervals
LASA study: Chair Stands Test | 21 years: 7 waves separated by 3 year intervals
LASA study: Walking Test | 21 years: 7 waves separated by 3 year intervals
LASA study: Cardigan Test | 21 years: 7 waves separated by 3 year intervals
LASA study: Balance Test | 21 years: 7 waves separated by 3 year intervals

OTHER OUTCOMES:
InterRAI: Cognitive Performance Scale | 16 months
InterRAI: ADL Hierarchy Scale | 16 months
InterRAI: Timed 4 meter Walk Test | 16 months
InterRAI: Distance walked in past 3 days | 16 months
InterRAI: Hours of physical activity in past 3 days | 16 months
InterRAI: Days of coming outside in past 3 days | 16 months

IPD SHARING:
Plan to Share IPD: Undecided
Not Applicable: Permission to use the data should be obtained from the LASA and/or InterRAI researchers